CLINICAL TRIAL: NCT04864691
Title: Department of Interventional Neurology, Beijing Tiantan Hospital, Capital Medical University
Brief Title: Endovascular Recanalization and Standard Medical Management for Symptomatic Nonacute Intracranial Artery Occlusion Trial
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Feng Gao (Other)
Responsible Party: Sponsor-Investigator, Feng Gao, Department of Interventional Neurology, Beijing Tiantan Hospital, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018AAA0102600
Record Dates: First submitted 2021-04-19; First posted 2021-04-29 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Intracranial Artery Occlusion With Infarction
Keywords: standard medical therapy; symptomatic non-acute intracranial artery occlusion; endovascular recanalization

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endovascular recanalization plus standard medical treatment (Experimental): patients with symptomatic non-acute intracranial artery occlusion treated by endovascular recanalization and standard medical treatment after procedure
  Interventions: Biological: endovascular recanalization
- standard medical treatment (Active Comparator): Patients take aspirin 100 mg/day or clopidogrel 75mg/day for the entire follow-up period (EVR patients take aspirin 100 mg/day and clopidogrel 75mg/day for 30-90 days after procedure)
  Interventions: Biological: endovascular recanalization

INTERVENTIONS:
Biological: endovascular recanalization — to recanalize the occlusion cerebral artery with intravascular intervention

SUMMARY:
Background The management of patients with symptomatic nonacute intracranial artery occlusion (sNA-ICAO), which is a special subset with high morbidity and a high probability of recurrent serious ischemic events despite standard medical therapy (SMT), has been clinically challenging. Some small-sample clinical studies have also discussed endovascular recanalization for sNA-ICAO; however, there is currently a lack of evidence from multicenter, prospective, large-sample cohort trials. The aim of our present study was to evaluate the technical feasibility and safety of endovascular recanalization for sNA-ICAO.

Methods and analysis: Our group is currently undertaking a multisite, nonrandomized cohort, prospective registry study enrolling consecutive patients presenting with sNA-ICAO at 15 centers in China between May 1, 2020, and April 30, 2023. A cohort of patients who received SMT and a cohort of similar patients who received ER plus SMT were constructed and followed up for 2 years. The primary outcome is the composite of stroke/TIA within 2 years following enrollment and stroke/TIA ipsilateral to the target vessel. The secondary efficacy outcome includes the following two parts: 1) the incidence of stroke/TIA ipsilateral to the target vessel within 30 days and 90 days in both groups; 2) the all-cause mortality, mRS score, NIHSS score and cognitive function at 30 days, 90 days, 8 months, 12 months and 24 months for both groups, including the MRI, CTA/MRA, CTP or MRP results in patients with internal carotid artery or middle cerebral artery occlusion as well as CTA in patients with basilar or vertebral artery occlusion at 90 days, 12 months and 24 months. Descriptive statistics and linear/logistic multiple regression models will be generated. Clinical relevance will be measured as relative risk reduction, absolute risk reduction and the number needed to treat.

Ethics and dissemination This study protocol was reviewed and approved primarily by Beijing Tiantan Hospital, the Capital Medical University Medical Ethics Committee, and the institutional review boards of all partner sites. The study is being externally monitored, and the results will be published in open-access peer-reviewed scientific journals and presented to academic and policy stakeholders.

ELIGIBILITY:
inclusion criteria:

1. Patient age ≥ 18 years old and life expectancy of 5 years or more.
2. Symptomatic sNA-ICAO defined as:diagnosed by CTA or MRA and confirmed by angiography; Vascular occlusion time more than 24 hours;TIA or ischemic stroke (confirmed by CT or MRI) related to the LCAO despite SMT < 90 days prior to enrollment.
3. Modified Rankin scale score 0-2 at the time of informed consent.
4. More than one risk factor for atherosclerosis.
5. For patients with ICA or MCA M1 segment occlusion, ipsilateral hypoperfusion confirmed by CTP or MRI perfusion imaging prior to enrollment and analysis by the RAPID system.
6. For patients with intracranial segment occlusion of the vertebral artery, severe stenosis or occlusion of the contralateral vertebral artery.
7. Among women, no childbearing potential; or if a woman with childbearing potential, a negative pregnancy test result prior to randomization.
8. Agreement of the patient to comply with all protocol-specified follow-up appointments.
9. Signature by a patient of a consent form that has been approved by the local governing institutional review board (IRB)/medical ethics committee (MEC) of the respective clinical site.

exclusion criteria:

1. Intolerance or allergic reaction to a study medication without a suitable management alternative.
2. No atherosclerotic intracranial vasculopathies, such as dissection, moyamoya disease and vasculitis.
3. Concomitant intracranial aneurysms or any bleeding disorder.
4. Life expectancy <1 year due to other medical conditions.
5. Large infarction core, defined as an ASPECTS < 6 in anterior circulation and pc-ASPECTS < 6 points in posterior circulation.
6. For patients with MCA M1 segment occlusion, concomitant ≥50% stenosis of the proximal internal carotid artery or other intracranial arteries.
7. For patients with intracranial segment occlusion of the vertebral artery, continuance of the occluded vertebral artery to the posterior inferior cerebellar artery with no stump.
8. Incomplete clinical and imaging data.
9. Coexistent cardioembolic source (e.g., atrial fibrillation, mitral stenosis, prosthetic valve, MI within six weeks, intracardiac clot, ventricular aneurysm and bacterial endocarditis).
10. Occlusive lesions with severe calcification.
11. Platelet count <100,000/ml or history of heparin-induced thrombocytopenia.
12. Left ventricular ejection fraction <30% or admission for heart failure in the prior 6 months.
13. Extreme morbid obesity that would compromise patient safety during the procedure or the periprocedural period.
14. Coronary artery disease with two or more proximal or major diseased coronary arteries with 70% stenosis that have not or cannot be revascularized.
15. Anticoagulation with Marcumar, warfarin or direct thrombin inhibitors or anti-XA drugs.
16. Chronic atrial fibrillation.
17. Any history of atrial fibrillation or paroxysmal atrial fibrillation in the past 6 months that is considered to require long-term anticoagulant therapy.
18. Other high-risk cardiogenic embolisms, including left ventricular aneurysm, severe cardiomyopathy, aortic or mitral mechanical heart valve, severe calcified aortic stenosis (valve area < 1.0 cm2), endocarditis, moderate to severe mitral stenosis, left atrial thrombus or any intracardiac mass or known paradoxical embolism of unrepaired PFO.
19. Unstable angina defined as rest angina with ECG changes that is not amenable to revascularization (patients should undergo planned coronary revascularization at least 30 days before randomization).
20. Any major surgery, major trauma, revascularization procedure or acute coronary syndrome within the past 1 month.
21. serum creatinine >2.5 mg/dl or estimated GFR <30 cc/min.
22. Major surgery planned within 3 months after enrollment.
23. Currently listed or being evaluated for major organ transplantation (i.e., heart, lung, liver and kidney).
24. Participation in other trials and may affect the results of this study.
25. Inability to understand and cooperate with research procedures or provide informed consent.
26. Endarterectomy, bypass or stent implantation performed on the proximal end of the occlusion vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: feng feng, professor, Study Chair — Beijing Tiantan Hospital
Locations (15):
- China (15):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Beijing You 'anmen Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Liangxiang Hospital, Beijing, Beijing Municipality
  - Handan Central Hospital, Handan, Hebei
  - Hebei Provincial People's Hospital, Shijiazhuang, Hebei
  - ORDOS Central Hospital, Ordos, Inner Mongolia
  - TongLiao City Hospital, Tongliao, Inner Mongolia
  - Jingjiang people's Hospital, Jingjiang, Jiangsu
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - Tai'an Hospital of Traditional Chinese Medicine, Tai’an, Shandong
  - Tong Ren Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Taiyuan Central Hospital, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Taizhou first people's Hospital, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Zhang H, Han J, Sun X, Miao Z, Guo X, Xu G, Sun Y, Wen C, Wang C, Wu Y, Xu Y, Jiang Y, Zhang S, Liu C, Li D, Liu Y, Xu C, Gao F. Endovascular Recanalization and Standard Medical Management for Symptomatic Non-acute Intracranial Artery Occlusion: Study Protocol for a Non-randomized, 24-Month, Multicenter Study. Front Neurol. 2021 Sep 28;12:729534. doi: 10.3389/fneur.2021.729534. eCollection 2021. PMID 34650509

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endovascular Recanalization Plus Standard Medical Treatment | Standard Medical Treatment
Started | 154 | 299
Completed | 148 | 288
Not Completed | 6 | 11

BASELINE CHARACTERISTICS:
Population: 17 patients lost to 1 year follow-up
Groups:
- Total: Total of all reporting groups
Arm/Group | Endovascular Recanalization Plus Standard Medical Treatment | Standard Medical Treatment | Total
Number analyzed (Participants) | 154 | 299 | 453
Age, Categorical [Count of Participants; unit: Participants] — Baseline age of patients Population: 17 patients lost to 1 year follow-up
  Participants
    number analyzed (Participants) | 148 | 288 | 436
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 113 | 207 | 320
    >=65 years | 35 | 81 | 116
Age, Continuous [Mean (Inter-Quartile Range); unit: years] — Population: 17 patients lost to 1 year follow-up
  years
    number analyzed (Participants) | 148 | 288 | 436
    (all) | 57 [49 to 64] | 58 [50 to 65] | 57 [50 to 65]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 17 patients lost to 1 year follow-up
  Participants
    number analyzed (Participants) | 148 | 288 | 436
    Female | 42 | 72 | 114
    Male | 106 | 216 | 322
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 154 | 299 | 453
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome
Description: The primary outcome was a composite of any stroke or death within 30 days after enrollment or ischemic stroke in the territory of the qualifying artery from 30 days to 1 year after enrollment.
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Recanalization Plus Standard Medical Treatment | Standard Medical Treatment
Number analyzed (Participants) | 148 | 288
Participants | 27 | 21

2. Secondary Outcome: Incidence of Stroke/ TIA Ipsilateral to the Target Vessel
Description: stroke/ TIA ipsilateral to the target vessel will be defined according to the World
Time Frame: within 30 days and 90 days in both groups
Reporting Status: Not Posted

3. Secondary Outcome: All-cause Mortality, mRS Score, NIHSS Score and Cognitive Function
Description: to evaluate the change in all-cause mortality, mRS score, NIHSS score and cognitive function in the two groups
Time Frame: t 30 days, 90 days, 8 months, 12 months and 24 months for both groups
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Endovascular Recanalization Plus Standard Medical Treatment | Standard Medical Treatment
All-Cause Mortality (participants affected / at risk) | 7/148 | 5/288
Serious Adverse Events (participants affected / at risk) | 9/148 | 0/288
Other Adverse Events (participants affected / at risk) | 0/148 | 0/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Endovascular Recanalization Plus Standard Medical Treatment (N=148) | Standard Medical Treatment (N=288)
Serious Adverse Event (Vascular disorders) | 9 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT04864691/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT04864691/SAP_001.pdf